CLINICAL TRIAL: NCT04587674
Title: Identification of Outcome Predictors and Stratification of Responder Profiles Implanted With Spinal Cord Stimulation. An AI-based-pathway & Algorithmic Approach to Treat Failed Back Surgery Syndrome Patients
Acronym: PREDIBACK 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-A01734-35
Record Dates: First submitted 2020-09-04; First posted 2020-10-14 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pain, Intractable
MeSH Terms: conditions — Pain, Intractable | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spinal Cord Stimulation (Other)
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Lead(s) and Implant Pulse Generator

SUMMARY:
Failed Back Surgery Syndrome is commonly defined as new, recurrent, or persistent pain in the back and/or leg(s) of at least 6-month duration following spinal surgery. The literature estimates that 10-50% of patients undergoing spinal surgery are likely to develop such pain, representing a substantial financial burden. Among them, 5-10% would suffer from severe pain, which are intense, neuropathic and generally refractory to conventional therapeutic strategies considerably affect patients' functional capacity as well as their psychological and social well-being.

Spinal Cord Stimulation (SCS) is a well-established therapy to alleviate severe intractable neuropathic pain such as FBSS. SCS is a safe and reversible treatment option, which leads to improvement in pain relief and quality of life for patients with FBSS. Despite encouraging results in a chronic painful patient population that is refractory to conventional therapies, the literature estimates that only 58% [53% - 64%] of patients implanted with SCS devices achieved adequate pain relief.

FBSS population characterization and stratification and predictive modeling of SCS outcome are thus crucial to delineate future treatment options and to deliver neuromodulation therapy to the right patient.

The investigators designed a clinical prospective project based on SCS outcome optimization and SCS candidates' stratification: PREDIBACK 2.

This study would be a following part of a continuous project (PREDIBACK) that aims to better understand and stratify the therapies (drugs, surgery, psychological therapy or SCS) proposed to FBSS patients. The goal of PREDIBACK 1 was to develop a decision tool that simplifies the therapeutic decision process.

PREDIBACK 2 will focus on the neuromodulation pathway. Easing and helping patient orientation should improve referral yielding to specialists and accelerate patient flow through care pathway. Hence, facilitating access to adequate therapies for FBSS patients who usually have a longstanding history of pain.

ELIGIBILITY:
Selection Criteria:

* Subject is ≥ 18 years and ≤ 80 years.
* Subject has FBSS and does not require further surgery. For the purpose of this study, FBSS is defined as persistent or recurrent low back and leg pain of at least 6-month duration following at least one decompression and/or fusion procedure.
* Subject has persistent low back and leg pain despite other treatment modalities (pharmacological, surgical, physical, or psychological therapies) that have been tried and did not prove satisfactory or are unsuitable or contraindicated for the subject.
* VAS global pain is ≥ 50 mm.
* Subject meets the criteria for spinal cord stimulation test according to HAS guidelines (multidisciplinary consultation, psychological assessment...).
* Absence of active psychosis or history of serious psychotic illness requiring hospitalization.
* Subject understands and accepts the constraints of the study.
* Patient covered by French national health insurance.
* Patient who has given written consent to the study after having received clear information.

Non-inclusion Criteria:

* Subject is or has been treated with SCS, subcutaneous or peripheral nerve stimulation, an intrathecal drug delivery system, requires back surgery at the localization related to his/her original back pain complaint or experimental therapies.
* Subject low back pain is coming from a non-FBSS etiology (i.e. cancerous pain, infectious disease, etc.).
* Cause of low back pain accessible to etiological "mechanical" surgical treatment (discogenic low back pain, vertebral instability, spinal deformity, etc.).
* Subject had most recent back surgery less than 6 months ago.
* Simultaneous participation to any interventional study during the study
* Subject requiring closer protection, i.e. minors, pregnant women, nursing mothers, subjects deprived of their freedom by a court or administrative decision, subjects admitted to a health or social welfare establishment, major subjects under legal protection, and finally patient in an emergency setting.

  * MRI contraindications if MRI is not available within a time frame of 2 years from the last spinal surgery. Absolute contraindications are: Cardiac implantable electronic device, metallic intraocular foreign bodies, cochlear implants, drug infusion pumps, catheters with metallic components, cerebral artery aneurysm clips, magnetic dental implants, tissue expander, artificial limb, hearing aid, piercing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Composite SCS efficacy score | 6 months
  Rate of SCS responders is defined as having at least three of these criteria:
  * Having at least a 30% decrease in Oswestry Disability Index (ODI) percentage. 10 items ranging from 0 to 5 where 0 indicates high ability and 5 indicate the inability.
  * Having at least a 50% decrease in the Visual Analogic Scale (VAS) (0 = no back pain, 10=worst imaginable pain)
  * Having at least a 0.2 points increase in the EuroQol-5 Dimensions (EQ-5D) questionnaire score. The maximum score of 1 indicates the best possible quality of life.
  * Having a decrease of 1.4 points in the Hospital Anxiety-Depression Scale (HADS) score. The total score ranges from 0 to 24 for each category.
  * 30% decrease pain surface (cm²): pain will assess painful area in terms of intensity, surface and pain typology.
  * Having a Patient Global Impression of Change (PGIC) score of at least 6. PGIC is a 7-point scale.
  * Drug intake will be measured using the Medication Quantification Scale (MQS) with a reduction of 3.4 points.

SECONDARY OUTCOMES:
Pain intensity | 6 months
  Pain intensity will be assessed using the Visual Analogic Scale (VAS score : 0 "no pain" to 10 "worst pain")
Pain surface | 6 months
  Pain mapping criteria will be compared. Pain mapping criteria include: Global Pain Surface (cm²), Pain intensities associated with the surface measurements, Mechanical/neuropathic components of pain surfaces.
Functional capacity | 6 months
  Functional capacity will be assessed using the Oswestry Disability Index (ODI, 0 "no disability" to 100% "complete disability")
Impact of Quality of life | 6 months
  Quality of life will be assessed using the EuroQol Five Dimensions index (EQ5D, 0 "dead" to 1 "perfect health")
Psychological distress | 6 months
  Psychological distress will be assessed using the Hospital Anxiety and Depression Scale (HADS, For each subscale the total score is at most 21. A score of ≥11 is considered a clinically significant disorder)
Social insecurity | 6 months
  Social insecurity will be assessed using the EPICES questionnaire [0 = low risk of insecurity to 100 = high risk of insecurity]
Psychological resilience | 6 months
  Psychological resilience will be assessed using the CD-RISC-10 (10-item Connor-Davidson Resilience Scale) questionnaire. [0 = low resilience to 40 = high resilience]
Effects of the technical parameters and Spinal Cord Stimulation devices on paresthesia | 6 months
  % of Type of lead (Spinal Cord Stimulation Monocolumn vs Multicolumn Lead)
Effects of the technical parameters and Spinal Cord Stimulation devices on paresthesia | 6 months
  Stimulation intensity (mA, milliAmper)
Effects of the technical parameters and Spinal Cord Stimulation devices on paresthesia | 6 months
  Stimulation pulse width (µs, microsecond)
Effects of the technical parameters and Spinal Cord Stimulation devices on paresthesia | 6 months
  Stimulation frequency (Hz, Hertz)
Effects of the technical parameters and Spinal Cord Stimulation devices on paresthesia | 6 months
  % of Stimulation Waveform (Low Dose, High Dose, Both), Electrical parameters
Spinal Cord Stimulation efficacy using objective measurement tools | 6 months
  Intellis/SnapshotTM platform to the ActiGraph GT9X.
  -Duration of standing position given by both Intellis and GT9X,
Spinal Cord Stimulation efficacy using objective measurement tools | 6 months
  Intellis/SnapshotTM platform to the ActiGraph GT9X.
  -Duration of sitting position given by both Intellis and GT9X,
Spinal Cord Stimulation efficacy using objective measurement tools | 6 months
  Intellis/SnapshotTM platform to the ActiGraph GT9X.
  -Duration of lying position given by both Intellis and GT9X,
Spinal Cord Stimulation efficacy using objective measurement tools | 6 months
  Intellis/SnapshotTM platform to the ActiGraph GT9X.
  -Duration of mobile position (activity) given by both Intellis and GT9X,
Spinal Cord Stimulation efficacy using objective measurement tools | 6 months
  Intellis/SnapshotTM platform to the ActiGraph GT9X.
  -Number of steps given by GT9X,
Spinal Cord Stimulation efficacy using objective measurement tools | 6 months
  Intellis/SnapshotTM platform to the ActiGraph GT9X.
  -Sleep duration given by GT9X,
Spinal Cord Stimulation efficacy using objective measurement tools | 6 months
  Intellis/SnapshotTM platform to the ActiGraph GT9X.
  -Sleep efficacy given by GT9X,
Spinal Cord Stimulation efficacy using objective measurement tools | 6 months
  Intellis/SnapshotTM platform to the ActiGraph GT9X.
  -Sleep onset latency given by GT9X,

CONTACTS AND LOCATIONS:
Overall Officials: Philippe RIGOARD, MD, PhD, Principal Investigator — Poitiers Hospital University
Locations (7):
- France (7):
  - Caen Univerisity Hospital, Caen
  - Parc Polyclinic, Caen
  - Louis Pasteur Hospital, Colmar
  - Lyon University Hospitals, Lyon
  - Nice University Hospital, Cimiez Hospital, Nice
  - Poitiers Hospital University, Poitiers
  - Foch Hospital, Suresnes

IPD SHARING:
Plan to Share IPD: No